CLINICAL TRIAL: NCT02553707
Title: Open-Label Study to Establish the Short Term Efficacy of Intravenous Loading-Doses of Bondronat 6 mg in Patients With Breast Cancer and Skeletal Metastases Experiencing Moderate to Severe Pain, Within 7 Days After Initiation of Treatment
Brief Title: A Study to Assess the Short Term Efficacy of Intravenous Ibandronate (Bondronat) in Participants With Metastatic Bone Pain Due to Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20268
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Pain; Bone Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Pain; Bone Neoplasms; Neoplasm Metastasis | interventions — Ibandronic Acid

ARMS (1):
- Ibandronate (Experimental): Participants will receive ibandronate 6 mg IV on Days 1, 2, and 3.
  Interventions: Drug: Ibandronate

INTERVENTIONS:
Drug: Ibandronate — Participants will receive ibandronate 6 mg IV on Days 1, 2, and 3.
  Other Names: Bondronat

SUMMARY:
This study will assess the short term efficacy of ibandronate (6 mg intravenous [IV]) in participants with breast cancer and malignant bone disease, with moderate to severe pain. All participants will receive an IV infusion of ibandronate on Days 1, 2, and 3, and pain response will be measured on Days 1-7. The anticipated time on study treatment is 3 days, and the target sample size is 182 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Female participants greater than or equal to (>=) 18 years of age
* Breast cancer with bone metastases
* Pain score of >=4 on Worst Pain scale of Brief Pain Inventory (BPI)
* Stable analgesic regimen.

Exclusion Criteria:

* Participants who have received a bisphosphonate within 3 weeks of start of trial
* Radiotherapy to bone within 4 weeks of enrolment
* Hypersensitivity to ibandronate
* Central nervous system (CNS) or meningeal metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with >=25% reduction in mean pain | up to Day 6
Percentage of participants with =<35% increase in mean analgesic consumption | up to Days 7

SECONDARY OUTCOMES:
Change from Baseline in average pain score | Baseline (Days 0), 5, and 7
Analgesic consumption | up to Day 7
Pain response | up to Day 7
Time to pain response | up to Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (10):
- Hungary (10):
  - Budapest
  - Győr
  - Gyula
  - Kecskemét
  - Nyíregyháza
  - Szeged
  - Székesfehérvár
  - Szombathely
  - Veszprém
  - Zalaegerszeg